CLINICAL TRIAL: NCT06234280
Title: Korean Multicenter Registry of ELUVIA Stent for Femoropopliteal Artery Disease
Acronym: K-ELUVIA
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2017-0095
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Symptomatic Peripheral Artery Disease With Femoropopliteal Lesions; Moderate or Severe Claudication (Rutherford Category 2 or 3); Critical Limb Ischemia (Rutherford Category 4 or 5)
Keywords: Peripheral artery disease; femoropopliteal; drug-eluting stent; restenosis
MeSH Terms: conditions — Lymphoma, Follicular; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eluvia: Patients treated with Eluvia stent
  Interventions: Device: Implantation of Eluvia stent

INTERVENTIONS:
Device: Implantation of Eluvia stent — Implantation of Eluvia stent

SUMMARY:
* Prospective, multi-center single-arm observational study
* A total of 100 subjects with femoropopliteal artery disease who meet all inclusion and exclusion criteria will be included.
* Patients will be followed clinically for 24 months after the procedure.
* An imaging study (duplex ultrasound, CT or catheter-based angiography) follow-up according to participating hospital's protocol will be performed at 12 months.
* Ankle-brachial index, symptom status and presence of stent fracture will be evaluated at 12 months.

DETAILED DESCRIPTION:
• Prospective, multi-center single-arm observational study

Screening (day 0):

1. Medical history and demography of the patient reviewed
2. Inclusion/exclusion eligibility will be checked
3. Physical examination (Height, weight)
4. Laboratory test

   * BUN, eGFR, Cr.
   * Hb, WBC, platelet
   * Lipid level (total cholesterol, LDL-C, triglyceride, HDL-C)
5. Ankle-brachial index
6. Imaging study (CT/MR angiography, Doppler ultrasound, or catheter angiography)
7. Medication

Enrollment (day 0):

1) Written consent

Post PTA (Day 1 ~3):

1. Adverse event
2. Ankle-brachial index
3. Laboratory test:

   * BUN, eGFR, Cr.
   * Hb, WBC, platelet
4. Concomitant medication Regular Follow-up Visits Visit 1 (post-PTA 30±14 days)

1) Symptom: Rutherford class 2) Laboratory test:

* BUN, eGFR, Cr.
* Hb, WBC, platelet 3) Concomitant medication 4) Adverse event Visit 2 (post-PTA 6 months ± 30 days)

  1. Symptoms: Rutherford class
  2. Ankle-brachial index
  3. Concomitant medication
  4. Adverse event Visit 3 (post-PTA 12 months ± 60 days)

  <!-- -->

  1. Symptoms: Rutherford class
  2. Ankle-brachial index
  3. Duplex ultrasound, CT, or catheter angiography
  4. Biplane radiograph of femur for evaluation of stent fracture
  5. Laboratory test
* BUN, eGFR, Cr.
* Hb, WBC, platelet
* Lipid level (total cholesterol, LDL-C, triglyceride, HDL-C) 6)Concomitant medication 7) Adverse event Visit4 (post-PTA 24 months ± 60 days)

  1. Symptom: Rutherford category
  2. Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years of older
2. Symptomatic peripheral artery disease:

   * Moderate or severe claudication (Rutherford category 2 or 3)
   * Critical limb ischemia (Rutherford category 4-5)
3. Femoropopliteal artery lesions with stenosis > 50%
4. ABI < 0.9 before treatment
5. Patents treated with ELUVIA stent for femoropopliteal artery disease
6. Patients with signed informed consent

Exclusion Criteria:

1. Acute critical limb ischemia
2. Severe critical limb ischemia (Rutherford category 6)
3. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, cilostazol, or contrast agents
4. In-stent restenosis lesions (Restenosis lesions without previously implanted stents are eligible to the enrollment)
5. Bypass graft lesions
6. Age > 85 years
7. Severe hepatic dysfunction (> 3 times normal reference values)
8. Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
9. LVEF < 40% or clinically overt congestive heart failure
10. Pregnant women or women with potential childbearing
11. Life expectancy <1 year due to comorbidity
12. Untreated proximal inflow disease of the ipsilateral iliac arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic peripheral artery disease with femoropopliteal lesions:
  * Moderate or severe claudication (Rutherford category 2 or 3)
  * Critical limb ischemia (Rutherford category 4 or 5) Age: ≥19 years, but not older than 85 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical patency | at 24 months
  Freedom from symptom worsening, as indicated by an increase in Rutherford category accompanied by a ≥ 0.15 decrease in ABI or > 50% restenosis on imaging studies at 24 months.

SECONDARY OUTCOMES:
Ankle-brachial index | at 12 and 24 months
  Ankle-brachial index defined as the ratio of the blood pressure at the ankle to the blood pressure in the upper arm
Ruthford category | at 12 and 24 months
  Rutherford category - symptom status by Rutherford category
target lesion revascularization | at 12 and 24 months
  Target lesion revascularization - accumulative rate of repeat interventions or surgery for the treatment of symptomatic restenosis (>50% stenosis) in the target lesion
stent fracture rate | at 12 and 24 months
  stent fracture rate - incidence of stent fracture by radiographs or fluoroscopy in 2 different projections

CONTACTS AND LOCATIONS:
Overall Officials: Young-Guk Ko, MD, Principal Investigator — Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea